CLINICAL TRIAL: NCT05559645
Title: DZD9008 in Patients With Locally Advanced or Metastatic Non-Small Cell Lung Cancer (NSCLC) With EGFR Mutations: Cohort Study
Brief Title: Assessing an Oral EGFR Inhibitor, DZD9008 in Patients With Advanced Non-small Cell Lung Cancer(NSCLC) With EGFR Mutations (WU-KONG15)
Acronym: WU-KONG15
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Collaborators: Dizal (Jiangsu) Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Wang mengzhao, Chief Director of Department of Respiratory and Critical Care Medicine, Peking Union Medical College Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DZ2021E0006
Record Dates: First submitted 2022-07-30; First posted 2022-09-29 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Non Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- Cohort 1: EGFR sensitizing mutations, T790M neg (Experimental)
  Interventions: Drug: DZD9008
- Cohort 2: EGFR sensitizing mutations (Experimental)
  Interventions: Drug: DZD9008
- Cohort 3: EGFR uncommon mutations (Experimental)
  Interventions: Drug: DZD9008
- Cohort 4: EGFR Exon20ins (Experimental)
  Interventions: Drug: DZD9008
- Cohort 5: EGFR sensitizing mutations (Experimental)
  Interventions: Drug: DZD9008
- Cohort 6: EGFR sensitizing mutations,T790M pos (Experimental)
  Interventions: Drug: DZD9008
- Cohort 7: EGFR Exon20ins treatment naive (Experimental)
  Interventions: Drug: DZD9008

INTERVENTIONS:
Drug: DZD9008 — Daily dosing of DZD9008 200mg
  Arms: Cohort 1: EGFR sensitizing mutations, T790M neg; Cohort 2: EGFR sensitizing mutations; Cohort 3: EGFR uncommon mutations; Cohort 4: EGFR Exon20ins; Cohort 5: EGFR sensitizing mutations; Cohort 6: EGFR sensitizing mutations,T790M pos
Drug: DZD9008 — Daily dosing of DZD9008 300mg
  Arms: Cohort 7: EGFR Exon20ins treatment naive

SUMMARY:
This study is a single center cohort study to access the anti-tumor efficacy, safety and tolerability of DZD9008 in patients with locally advanced or metastatic non-small-cell lung cancer (NSCLC) harboring epidermal growth factor receptor (EGFR) sensitizing mutations and EGFR uncommon mutations who have progressed following standard TKI therapy, and in treatment naive patients with NSCLC harboring EGFR Exon20 insertion mutation and EGFR sensitizing mutations.

ELIGIBILITY:
Inclusion Criteria:

1. To provide a signed and dated, written informed consent.
2. Aged ≥ 18 years old
3. Histologically or cytologically confirmed locally advanced or metastatic NSCLC with documented EGFR mutations from a local laboratory
4. ECOG performance status 0-1.
5. Predicted life expectancy ≥ 12 weeks
6. Patient must have measurable disease according to RECIST 1.1.
7. Patient who has progressed or intolerant to standard therapy (except treatment naïve patients in Cohort 4 and Cohort 7: with EGFR Exon20ins; and in Cohort 5 with EGFR sensitizing mutation).
8. Patients with brain metastasis (BM) can be enrolled under the condition that BM is stable, neurologically asymptomatic and does not require corticosteroid treatment.
9. Adequate organ system function.

   * Absolute neutrophil count (ANC) ≥ 1.5 x 10^9/L
   * Platelets ≥ 100 x 10^9/L
   * Hemoglobin ≥ 9 g/dL
   * Total bilirubin ≤ 1.5 x ULN if no liver metastases or ≤ 3 x ULN in the presence of documented Gilbert's Syndrome (unconjugated hyperbilirubinemia) or liver metastases
   * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5 x ULN if no liver metastases or ≤ 5 x ULN with liver metastases
   * Creatinine ≤ 1.5 x ULN, concurrent with calculated or measured creatinine clearance ≥ 50 mL/min as calculated by the Cockcroft-Gault method or ≥ 50 mL/min in 24 hours
   * International normalized ratio (INR) ≤ 1.5 x ULN and activated partial thromboplastin time (APTT) ≤ 1.5 x ULN;
   * Serum amylase ≤ 1.5 x ULN and serum lipase ≤ 1.5 x ULN

Exclusion criteria:

1. Known history of bleeding diathesis.
2. Prior malignancy within 2 years requires active treatment.
3. Any unresolved toxicities from prior therapy greater than CTCAE grade 1 at the time of first administration.
4. History of stroke or intracranial haemorrhage within 6 months before the first administration.
5. Spinal cord compression or leptomeningeal metastasis.
6. As judged by the investigator, any evidence of severe or uncontrolled systemic diseases, which would jeopardize compliance with the protocol, or active infection including hepatitis B, hepatitis C and human immunodeficiency virus (HIV).
7. Any of the following cardiac criteria:

   * Mean resting corrected QT interval (QTcF) > 470 msec obtained from 3 electrocardiograms (ECGs);
   * Any clinically significant abnormalities in rhythm, conduction or morphology of resting ECG, e.g., complete left bundle branch block, third degree heart block, and second-degree heart block, PR interval > 250 msec.
   * Any factors that increase the risk of QTcF prolongation, such as heart failure, hypokalemia, congenital long QT syndrome, family history of long QT syndrome or unexplained sudden death under 40 years of age in first degree relatives or any concomitant medication known to prolong the QT interval.
   * Prior history of atrial fibrillation within 6 months of first administration of DZD9008, except prior drug treatment related and recovered.
8. Past medical history of interstitial lung disease, drug-induced interstitial lung disease, radiation pneumonitis which required steroid treatment, or any evidence of clinically active interstitial lung disease.
9. Refractory nausea and vomiting, chronic gastrointestinal diseases, inability to swallow the formulated product or previous significant bowel resection that would preclude adequate absorption of DZD9008.
10. History of hypersensitivity to active or inactive excipients of DZD9008 or drugs with a similar chemical structure or class to DZD9008.
11. Women who are pregnant or breast feeding.
12. Involvement in the planning and conduct of the study.
13. Judgment by the investigator that the patient should not participate in the study if the patient is unlikely to comply with study procedures, restrictions and requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2021-11-18 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | through study completion, an average of 1 year
  To assess anti-tumor activity of DZD9008 according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 by investigator

SECONDARY OUTCOMES:
Duration of Response (DoR) | through study completion, an average of 1 year
  To assess anti-tumor activity of DZD9008 according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 by investigator

OTHER OUTCOMES:
Disease Control rate (DCR) | through study completion, an average of 1 year
  To assess anti-tumor activity of DZD9008 according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 by investigator
Objective Response Rate (ORR) | through study completion, an average of 1 year
  To assess anti-tumor activity of DZD9008 according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 by investigator
Overall survival (OS) | through study completion, an average of 1 year
  To assess anti-tumor activity of DZD9008 according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 by investigator
Number of participants with adverse events (AEs) according to CTCAE 5.0 | From first dose until 28 days after the last dose
  To assess safety and tolerability of DZD9008 when given orally to patients with advanced NSCLC
Number of participants with clinically significant laboratory assessment abnormalities | From first dose until 30 days after the last dose
  To assess safety and tolerability of DZD9008 when given orally to patients with advanced NSCLC
Number of participants with clinically significant abnormal vital signs | From first dose until 30 days after the last dose
  To assess safety and tolerability of DZD9008 when given orally to patients with advanced NSCLC
Number of participants with clinically significant 12-lead electrocardiograms (ECGs) abnormalities | From first dose until 30 days after the last dose
  To assess safety and tolerability of DZD9008 when given orally to patients with advanced NSCLC

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Respiratory and Critical Care Medicine, Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No